CLINICAL TRIAL: NCT02786836
Title: 13C-Methacetin Breath Test for the Prediction of Outcome in in Acute Liver Injury or Acute Liver Failure
Brief Title: 13C-Methacetin Breath Test for the Prediction of Outcome in in ALI or ALF
Acronym: ALFSG-MBT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Medical University of South Carolina (Other); University of Michigan (Other); Meridian Bioscience, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Lee, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 122015-008; U01DK058369 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-06-01 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Acute Liver Failure
Keywords: acute liver failure; methacetin; breath test; severe acute liver injury; hepatic encephalopathy; ALFSG Registry; acetaminophen toxicity
MeSH Terms: conditions — Liver Failure, Acute; Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 13C-Methacetin Testing (Experimental): All patients enrolled into the ALFSG Registry with the duration of illness <26 weeks with (1) severe acute liver injury; International Normalized Ratio (INR) ≥2.0) and not related to acetaminophen overdose, with no evidence of hepatic encephalopathy (HE); and (2) acute liver failure; INR ≥1.5 with presence of any degree of HE will perform the Breath Test.
  Interventions: Drug: 13C-Methacetin

INTERVENTIONS:
Drug: 13C-Methacetin — The test substrate in this study, ¹³C-methacetin solution for single-use oral administration (75 mg in 150 ml purified water), is administered orally or via feeding tube, rapidly absorbed, exclusively metabolized by hepatic mixed function oxidase via O-demethylation, mainly by cytochrome P450 enzyme, subtype 1A2, into acetaminophen and formaldehyde. The formaldehyde is then transformed through two successive oxidative steps to ¹³carbon dioxide, the quantity of which is measured in exhaled breath as a ratio of 13C to 12C.
  The nasal or intubated breath sampling investigational device (ID) circuit continuously transports the breath sample from the patient to the BreathID® MCS device before and following administration of the 13C-methylacetanilide test substrate.
  Other Names: N-(4)-13Cmethoxyphenyl acetamide

SUMMARY:
The ALFSG-MBT protocol is for a multicenter, open label, non-randomized study to determine the value of Breath Identification® (BreathID®) N-(4-Methoxy-13C-phenyl)acetamide (13C-Methacetin) Breath Test System in predicting the outcome of patients diagnosed with severe acute liver injury that is not related to acetaminophen overdose or acute liver failure who meet inclusion/exclusion criteria.

Up to 200 evaluable patients will be enrolled. An evaluable patient is one who has completed one or more breath tests for at least 30 minutes after administration of the 13C-Methacetin solution (test substrate).

The Breath Test will be performed up to five times during the study period on all enrolled patients. The first Breath Test will be performed upon admission into the study (Day 1) and repeated on Days 2, 3, 5 and 7 provided no contra-indications are present. Each test continuously measures changes in the metabolism of the 13C-Methacetin in order to assess the improvement or deterioration in liver metabolic function about improvement or deterioration in liver metabolic function. If an enrolled non-APAP ALI or ALF patient receives a liver transplant, is discharged /transferred from the hospital or dies prior to Day 7, additional Breath Tests will not be performed.

Patients will be contacted for the Day 21 follow up (21 days after enrollment into the trial) to determine spontaneous survival, transplantation and occurrence of serious adverse events since the patient's last study treatment.

DETAILED DESCRIPTION:
The importance of identifying the patient with with ALI or ALF who is likely to die without a liver transplant cannot be overstated and has remained a primary focus of clinical investigation for 25 years. A recent analysis also conducted by the Acute Liver Failure Study Group (ALFSG) found that poor outcomes in the ALI patients are less frequent than is observed in the ALF population. However, in cases where ALI was not related to an acetaminophen (APAP) overdose, progression to poor outcomes was similar. Traditional scoring systems and prognostic models, such as King's College Criteria (KCC), Sequential Organ Failure Assessment (SOFA) and Acute Physiology and Chronic Health Evaluation II (APACHE II), currently used to monitor patients with ALF lack individual sensitivity and specificity and do not provide direct information about the liver's metabolic function, which is a key variable in assessing liver status and potential disease progression versus recovery in ALF patients. Despite recent advances used by the ALFSG Prognostic Index (ALFSG-PI), ALI Prognostic Index (ALI-PI) and Model for End-Stage Liver Disease (MELD), better predictive modalities are still needed.

The 13C-Methacetin breath test is a rapid, reproducible, point-of-care test of liver metabolic function. After oral or naso-enteric/orogastric tube administration, the 13C labeled Methacetin is O-demethylated by cytochrome P450 1A2 (liver enzyme name) in the liver and further biotransformed into carbon dioxide labeled with carbon 13 (13CO2), which is expired in breath. The BreathID® Molecular Correlation Spectroscopy (MCS) device captures and quantifies expired 13CO2 and standardizes recovery against expired normal carbon dioxide (12CO2) through a nasal cannula (in conscious patients) or an adaptor connected to the ventilator line (for intubated patients). The results obtained from the device are expressed as delta over baseline (DOB), which expresses the change in 13CO2/12CO2 ratio in comparison to the baseline measurement. It can be transformed into the percentage of 13C dose recovered over time (PDR) after the ingestion of Methacetin, and the cumulative PDR (CPDR), the rate at which 13C substrate is metabolized, derived from the breath 13C/12C ratio.

This is a multicenter, open label, non-randomized study of the MBT to assess functional trends of liver metabolism in patients diagnosed with severe acute liver injury not related to acetaminophen overdose (non-APAP ALI) or acute liver failure (ALF). Up to 200 evaluable patients with non-APAP ALI or ALF present at the time of enrollment into the ALFSG Registry will be consecutively enrolled. An evaluable patient is one who has completed one or more Breath Tests measured for a minimum of 30 (and ideally 60) minutes after administration of the 13C-Methacetin solution. Study sites will include up to 11 of the clinical sites located in the United States that are involved in the ALFSG.

The Breath Test will be performed up to five times during the study period on all enrolled subjects. The first Breath Test will be performed as close to the time of study enrollment as possible upon admission into the study (Day 1). The Breath Test will be repeated on Days 2, 3, 5 and 7 as close as possible to the same time of day as the first Breath Test. If a subject who is enrolled into the ALFSG-MBT Trial with non-APAP ALI converts to ALF, breath test collection will continue until a maximum of five Breath Tests have been performed. If an enrolled non-APAP ALI or ALF subject receives a liver transplant, is discharged/transferred from the hospital or dies prior to Day 7, no additional Breath Tests will be performed. Enrolled patients will be contacted for the Day 21 follow up (21 days after the subject's enrollment into the trial) to determine spontaneous survival, transplantation and occurrence of serious adverse events since the subject's last study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women (18-80 years of age)
2. Severe acute liver injury not related to acetaminophen overdose: INR ≥2.0; no evidence of HE
3. Acute liver failure: INR ≥1.5; presence of any degree of HE
4. Duration of illness <26 weeks
5. Enrolled into the ALFSG Registry.
6. Written informed consent from the patient or patient's legally authorized representative or family member as defined in the Federal Register Number 21 Congressional Federal Register (CFR)50.3(m)

Exclusion Criteria:

1. Evidence of pre-existing chronic liver disease
2. Pre-existing New York Heart Association stage III/IV heart failure
3. Evidence of pre-existing chronic renal failure
4. Chronic hemodialysis prior to hospital admission
5. Evidence of cirrhosis (unless clinically acute Wilson disease or autoimmune non-APAP ALI or ALF)
6. Severe obstructive lung disease (FEV1 <50% of predicted on previous spirometry)
7. Severe shock, defined as mean arterial pressure (MAP) <70 mmHg despite >15 µg/kg/min dopamine, >0.1 µg/kg/min epinephrine, or >0.1 norepinephrine µg/kg/min
8. Extensive small bowel resection (>50 cm)
9. Any evidence of upper GI bleeding at enrollment requiring intervention (endoscopy or red blood cell (RBC) transfusion specifically for upper GI bleeding)
10. Liver transplantation (LT) prior to enrollment. (Note: Listing for LT does not preclude participation in the trial.)
11. Pregnancy or breastfeeding women (Note: Pregnancy related non-APAP ALI or ALF may be considered for entry following the delivery of the baby and assuming the mother does not wish to breastfeed or collect breast milk during the study period.)
12. Allergic to acetaminophen (such as Tylenol® or any other acetaminophen-containing medications)
13. Participation in other clinical studies evaluating other experimental treatments or procedures. (Note: Participation in observatory studies is not an exclusion.)
14. Patients in whom enteral drugs or fluids are contra-indicated or the patient either does not have an appropriately placed naso-enteric/orogastric tube in situ or cannot tolerate taking the drug preparation orally (200 ml)
15. Budd-Chiari Syndrome
16. Non-APAP ALI or ALF caused by malignancy
17. Moderate and severe adult respiratory distress syndrome (ARDS), as defined by Berlin Criteria.
18. Subjects who have received amiodarone in the 30 days prior to study enrollment
19. Consumption of any food or beverage that contains caffeine in the 24 hours prior to enrollment
20. Consumption of any of the following drugs that may interfere with the metabolism of 13C-Methacetin in the 48 hours prior to study enrollment including: allopurinol, carbamazepine, cimetidine, ciprofloxacin, daidzein, disulfiram, Echinacea, enoxacin, fluvoxamine, methoxsalen, mexiletine, montelukast, norfloxacin, phenylpropanolamine, phenytoin, propafenone, rifampin, terbinafine, ticlopidine, thiabendazole, verapamil, zileuton or oral contraceptives
21. Consumption of alcohol in the 24 hours prior to enrollment
22. Smoking cigarettes in the 8 hours prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Fontana, MD, Study Chair — University of Michigan
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University Medical Center, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - VCU Medical Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data for the overall study will be shared once the study is completed.

REFERENCES:
- [Background] O'Grady JG, Alexander GJ, Hayllar KM, Williams R. Early indicators of prognosis in fulminant hepatic failure. Gastroenterology. 1989 Aug;97(2):439-45. doi: 10.1016/0016-5085(89)90081-4. PMID 2490426
- [Background] Cholongitas E, Senzolo M, Patch D, Kwong K, Nikolopoulou V, Leandro G, Shaw S, Burroughs AK. Risk factors, sequential organ failure assessment and model for end-stage liver disease scores for predicting short term mortality in cirrhotic patients admitted to intensive care unit. Aliment Pharmacol Ther. 2006 Apr 1;23(7):883-93. doi: 10.1111/j.1365-2036.2006.02842.x. PMID 16573791
- [Background] Craig DG, Ford AC, Hayes PC, Simpson KJ. Systematic review: prognostic tests of paracetamol-induced acute liver failure. Aliment Pharmacol Ther. 2010 May;31(10):1064-76. doi: 10.1111/j.1365-2036.2010.04279.x. Epub 2010 Feb 24. PMID 20180786
- [Background] Stravitz RT, Reuben A, Mizrahi M, Lalazar G, Brown K, Gordon SC, Ilan Y, Sanyal A. Use of the methacetin breath test to classify the risk of cirrhotic complications and mortality in patients evaluated/listed for liver transplantation. J Hepatol. 2015 Dec;63(6):1345-51. doi: 10.1016/j.jhep.2015.07.021. Epub 2015 Jul 26. PMID 26220750
- [Background] Lalazar G, Adar T, Ilan Y. Point-of-care continuous (13)C-methacetin breath test improves decision making in acute liver disease: results of a pilot clinical trial. World J Gastroenterol. 2009 Feb 28;15(8):966-72. doi: 10.3748/wjg.15.966. PMID 19248196
- [Background] Goetze O, Selzner N, Fruehauf H, Fried M, Gerlach T, Mullhaupt B. 13C-methacetin breath test as a quantitative liver function test in patients with chronic hepatitis C infection: continuous automatic molecular correlation spectroscopy compared to isotopic ratio mass spectrometry. Aliment Pharmacol Ther. 2007 Jul 15;26(2):305-11. doi: 10.1111/j.1365-2036.2007.03360.x. PMID 17593076
- [Background] Nista EC, Fini L, Armuzzi A, Candelli M, Zocco MA, Cazzato IA, Merra G, Finizio R, Miele L, Grieco A, Gasbarrini G, Gasbarrini A. 13C-breath tests in the study of microsomal liver function. Eur Rev Med Pharmacol Sci. 2004 Jan-Feb;8(1):33-46. PMID 15209153
- [Background] Starmer GA, McLean S, Thomas J. Analgesic potency and acute toxicity of substituted anilides and benzamides. Toxicol Appl Pharmacol. 1971 May;19(1):20-8. doi: 10.1016/0041-008x(71)90185-2. No abstract available. PMID 5570565
- [Background] de Franchis R. Updating consensus in portal hypertension: report of the Baveno III Consensus Workshop on definitions, methodology and therapeutic strategies in portal hypertension. J Hepatol. 2000 Nov;33(5):846-52. doi: 10.1016/s0168-8278(00)80320-7. No abstract available. PMID 11097497
- [Background] Lalazar G, Pappo O, Hershcovici T, Hadjaj T, Shubi M, Ohana H, Hemed N, Ilan Y. A continuous 13C methacetin breath test for noninvasive assessment of intrahepatic inflammation and fibrosis in patients with chronic HCV infection and normal ALT. J Viral Hepat. 2008 Oct;15(10):716-28. doi: 10.1111/j.1365-2893.2008.01007.x. Epub 2008 Jul 11. PMID 18638013
- [Background] Lalazar G, Mullhaupt, B., Margalit M. Point of care non-invasive 13C methacetin breath testing accurately identifies significant liver inflammation and fibrosis: a novel method for assessing liver damage. Gastroenterology; 2007 abstract
- [Background] Allman K, Wilson I. Oxford Handbook of Anaesthesia. 2nd ed. New York: Oxford University Press 2006;xxiv:1203.
- [Background] Lee WM, James L, Wendon J, Stravitz RT, Pop OT, Audimoolam VK. Does Methacetin breath testing increase acetaminophen hepatotoxicity in the setting of acute liver failure? Hepatology 2015: Accepted for poster presentation at the AASLD Liver Meeting held in San Francisco from November 13-17, 2015.
- [Background] Audimoolam VK, Patel VC, Bernal W, Meir M, Lalazar G, Ilan Y, Wendon J. Use of an on-line at the point of care 13C-methacetin breath test as an adjunct tool for decision making in patients with acute liver failure. Hepatology 56;4Suppl:970A.
- [Background] Koch DG, Battenhouse H, Durkalski V, Lee WM, Reuben A. Clinical predictors of spontaneous survival in acute liver failure (ALF) patients with advanced coma. Hepatology 56;4Suppl:964A.
- [Background] Koch DG, Speiser JL, Durkalski V, Fontana RJ, Davern T, McGuire B, Stravitz RT, Larson AM, Liou I, Fix O, Schilsky ML, McCashland T, Hay JE, Murray N, Shaikh OS, Ganger D, Zaman A, Han SB, Chung RT, Brown RS, Munoz S, Reddy KR, Rossaro L, Satyanarayana R, Hanje AJ, Olson J, Subramanian RM, Karvellas C, Hameed B, Sherker AH, Lee WM, Reuben A. The Natural History of Severe Acute Liver Injury. Am J Gastroenterol. 2017 Sep;112(9):1389-1396. doi: 10.1038/ajg.2017.98. Epub 2017 Apr 25. PMID 28440304
- [Derived] Stravitz RT, Fontana RJ, Karvellas C, Durkalski V, McGuire B, Rule JA, Tujios S, Lee WM; Acute Liver Failure Study Group. Future directions in acute liver failure. Hepatology. 2023 Oct 1;78(4):1266-1289. doi: 10.1097/HEP.0000000000000458. Epub 2023 May 16. PMID 37183883
- See also: Acute Liver Failure Study Website — http://www.utsouthwestern.edu/labs/acute-liver/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with acute liver failure (ALF) who were enrolled into the ALF Study Group Registry at 11 participating investigative U.S. sites were screened for eligibility. In March 2018, patients with acute liver injury (ALI) not related to acetaminophen overdose (APAP) and enrolled into the ALFSG Registry were included and screened for eligibility.
Groups:
- 13C-Methacetin Breath Test (MBT): For each MBT, a baseline measurement was taken for up to 15 minutes using a nasal cannula retrieval device for non-intubated patients or an airway adapter connection to the endotracheal tube of intubated patients that was connected to the Breath ID® molecular correlation spectrometry (MCS) device. After completion of the baseline segment, one 75 milligram (mg) dose of 13C-Methacetin (test substrate) mixed into 150 milliliters (ml) of water was orally ingested by non-intubated patients or administered via nasoenteric tube to intubated patients. The BreathID® MCS device measured expired 13CO2 (carbon-13 dioxide) over a period of up to 60 minutes. A maximum of 5 daily tests were administered on study days 1, 2, 3, 5 and 7 for up to 1 hour after test substrate administration. Patients were contacted 21 days following study enrollment to determine vital status and to check for the development of serious adverse events.
Period: Overall Study
Arm/Group | 13C-Methacetin Breath Test (MBT)
Started | 76
Eligible Patients Enrolled Into the Stud | 76
Completed | 62
Not Completed | 14
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 3
Not completed — Liver Transplantation | 2
Not completed — Device or Pharmacy Issues | 3

BASELINE CHARACTERISTICS:
Population: Eligible patients enrolled into the study with at least one 13C-MBT measured for a minimum of 30 minutes after ingestion of the 13C-Methacetin solution.
Groups:
- 13C-Methacetin Breath Test (MBT): For each MBT, a baseline measurement was taken for up to 15 minutes using a nasal cannula retrieval device for non-intubated patients or an airway adapter connection to the endotracheal tube of intubated patients that was connected to the Breath ID® MCS device. After completion of the baseline segment, one 75 mg dose of 13C-Methacetin (test substrate) mixed into 150 ml of water was orally ingested by non-intubated patients or administered via nasoenteric tube to intubated patients. The BreathID® MCS device measured expired 13CO2 over a period of up to 60 minutes. A maximum of 5 daily tests were administered on study days 1, 2, 3, 5 and 7 for up to 1 hour after test substrate administration. Patients were contacted 21 days following study enrollment to determine vital status and to check for the development of serious adverse events.
Arm/Group | 13C-Methacetin Breath Test (MBT)
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 43 [28 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49
  Black | 11
  Asian | 2
  Hispanic | 4
Day 1 MBT measured for a minimum of 30 minutes after ingestion of the 13C-Methacetin solution [Count of Participants; unit: Participants] | 56

OUTCOME MEASURES:

1. Primary Outcome: Peak Percent Dose Recovery (PDR) Value
Description: Peak PDR is the maximal percent dose recovery (PDR) rate which reflects the maximum rate of metabolism of 13C-methacetin measured as the change in 13CO2 / 12CO2 (normal carbon dioxide) ratio after ingestion of 13C-methacetin normalized using the patient's height and weight. The distributions of mean PDR Peak values were compared between TFS (transplant free survival) and non-TFS (death/transplant) at Day 21.
Time Frame: Days 1 and 21
Population: Eligible patients enrolled into the study with available Day 1 13C-MBT results and 21-day outcome.
Measure: Mean (Standard Deviation); unit: percentage per hour
Groups:
- 13C-Methacetin Breath Test (MBT): For each MBT, a baseline measurement was taken for up to 15 minutes using a nasal cannula retrieval device for non-intubated patients or an airway adapter connection to the endotracheal tube of intubated patients that was connected to the Breath ID® MCS device. After completion of the baseline segment, one 75 mg dose of 13C-Methacetin (test substrate) mixed into 150 ml of water was orally ingested by non-intubated patients or administered via nasoenteric tube to intubated patients. The BreathID® MCS device measured expired 13CO2 over a period of up to 60 minutes.
Arm/Group | 13C-Methacetin Breath Test (MBT)
Number analyzed (Participants) | 35
percentage per hour
  Mean Peak PDR for TFS subjects at Day 21: number analyzed (Participants) | 23
  Mean Peak PDR for TFS subjects at Day 21 | 10.2 (7.8)
  Mean Peak PDR for non-TFS subjects at Day 21: number analyzed (Participants) | 12
  Mean Peak PDR for non-TFS subjects at Day 21 | 1.9 (0.6)

2. Secondary Outcome: Peak Percent Dose Recovery (PDR) Value
Description: This outcome is similar to the peak PDR defined in the primary outcome but as a secondary we are looking at Day 1 or Day 2 peak PDR values. Peak PDR is the maximal percent dose recovery (PDR) rate which reflects the maximum rate of metabolism of 13C-methacetin measured as the change in 13CO2 / 12CO2 ratio after ingestion of 13C-methacetin normalized using the patient's height and weight. The distributions of mean PDR Peak values were compared between TFS and non-TFS (death/transplant) at Day 21.
Time Frame: The first MBT reading either on Day 1 or Day 2 and Day 21
Population: Eligible patients enrolled into the study with available Day 1 or Day 2 13C-MBT results and 21-day outcome.
Measure: Mean (Standard Deviation); unit: percentage per hour
Groups:
- 13C-Methacetin Breath Test (MBT): For each MBT, a baseline measurement was taken for up to 15 minutes using a nasal cannula retrieval device for non-intubated patients or an airway adapter connection to the endotracheal tube of intubated patients that was connected to the Breath ID® MCS device. After completion of the baseline segment, one 75 mg dose of 13C-Methacetin (test substrate) mixed into 150 ml of water was orally ingested by non-intubated patients or administered via nasoenteric tube to intubated patients. The BreathID® MCS device measured expired 13CO2 over a period of up to 60 minutes. A maximum of 5 daily tests were administered on study days 1, 2, 3, 5 and 7 up to 1 hour after test substrate administration. Patients were contacted 21 days following study enrollment to determine vital status and to check for the development of serious adverse events.
Arm/Group | 13C-Methacetin Breath Test (MBT)
Number analyzed (Participants) | 56
percentage per hour
  Day 1 or 2 MBT & Day 21 TFS: number analyzed (Participants) | 35
  Day 1 or 2 MBT & Day 21 TFS | 9.1 (6.8)
  Day 1 or 2 MBT & Day 21 non-TFS: number analyzed (Participants) | 21
  Day 1 or 2 MBT & Day 21 non-TFS | 2.3 (0.9)

3. Secondary Outcome: Cumulative Percent Dose Recovery 20 (cPDR20) Value
Description: The relationship between the cPDR (cumulative PDR of metabolized 13C-Methacetin 20 minutes after ingestion) in single time points of MBT measurements and TFS and non-TFS (death/transplant) at Day 21.
Time Frame: The first MBT reading either on Day 1 or Day 2 and Day 21
Population: Eligible patients enrolled into the study with the initial 13C-MBT conducted on Day 1 or Day 2, and 21 day outcome.
Measure: Mean (Standard Deviation); unit: percentage per hour
Arm/Group | 13C-Methacetin Breath Test (MBT)
Number analyzed (Participants) | 56
percentage per hour
  Day 1 or 2 MBT/transplant free survival at Day 21: number analyzed (Participants) | 35
  Day 1 or 2 MBT/transplant free survival at Day 21 | 1.4 (1.3)
  Day 1 or 2 MBT & Day 21 non-TFS: number analyzed (Participants) | 21
  Day 1 or 2 MBT & Day 21 non-TFS | 0.2 (.2)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE), suspected adverse reactions (SAR) and unanticipated adverse device effects (UADE) were collected from the initiation of the first MBT through study completion (e.g. Day 21, death, liver transplant or withdrawal of consent). Non-serious adverse events (AE) and adverse device effects (ADE) were collected from from the initiation of the first MBT through Day 7.
Description: ADEs caused by insufficiencies/inadequacies in instructions for use, deployment, implantation, installation, operation, investigational medical device malfunction, and event as a result of user error or intentional misuse. UADEs caused by/associated with a device, if effect, problem, or death was not previously identified in nature, severity, or degree of incidence in investigational plan/application on health/safety; life-threatening; or problem related to subject rights, safety, or welfare.
Arm/Group | 13C-Methacetin Breath Test (MBT)
All-Cause Mortality (participants affected / at risk) | 11/62
Serious Adverse Events (participants affected / at risk) | 28/62
Other Adverse Events (participants affected / at risk) | 40/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13C-Methacetin Breath Test (MBT) (N=62)
Acute hepatic failure (Hepatobiliary disorders) | 14 (14)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Brain injury (Nervous system disorders) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 7 (7)
Presyncope (Nervous system disorders) | 1 (1)
Transplant (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 13C-Methacetin Breath Test (MBT) (N=62)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Haemophilus infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Recruitment goal of 200 patients not met due to challenges including multiple concomitant contraindicated meds, fasting requirement, establishing rapport with patients' family members due to sudden nature of illness and concerns for liver transplant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT02786836/Prot_SAP_001.pdf